CLINICAL TRIAL: NCT07367815
Title: Allogeneic Intraveinous Injection of Adipose Tissue Derived-mesenchymal Stem Cells in Mild to Moderate Alzheimer Disease: a Phase I/II Trial
Brief Title: Allogeneic Adipose Tissue Derived-stem Cells in Alzheimer Disease
Acronym: A3D
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RC31/19/0501; 2022-502846-28-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-09; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease,; phase I/II,; safety,; mesenchymal stem cell,; adipose tissue
MeSH Terms: conditions — Alzheimer Disease | interventions — Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 50 millions AdMSC dose (Experimental): Allogeneic AdMSC (CellREADY® drug product), intravenous administration, dose of 50x106 or 100x106 AdMSC (from 3 to 6 patients, "50x106 AdMSC " group, group 1)
  Interventions: Drug: CellREADY® drug product IV dose of 50 millions; Diagnostic Test: cerebral RMI; Diagnostic Test: PET scan
- 100 millions AdMSc dose (Experimental): Allogeneic AdMSC (CellREADY® drug product), intravenous administration, dose of 50x106 or 100x106 AdMSC (from 3 to 6 patients, "100x106 AdMSC " group, group 2) if safety analysis of group 1 is correct.
  Interventions: Drug: CellREADY® drug product IV dose of 100 millions; Diagnostic Test: cerebral RMI; Diagnostic Test: PET scan

INTERVENTIONS:
Drug: CellREADY® drug product IV dose of 50 millions — Allogeneic AdMSC (CellREADY® drug product), intravenous administration, dose of 50 millions.
  Initially, 3 patients will receive the lowest dose (50x106 AdMSC). If the safety analysis of the first 3 patients infused at dose 50x106 AdMSC does not show clinically significant AEs after 6 months of follow-up, 100x106 AdMSC administration may be started in 3 new patients. On the other hand, if safety analysis of the first 3 patients shows a clinically significant AE, 3 new patients will be injected at this same dose before making a final decision on the possibility of dose escalation. Thus, the "100x106 AdMSC " group will only start after the 6-month follow-up and safety analysis completed in the "50x106 AdMSC " group. For each dose, all patients will be followed for 6 months post-injection with 6 visits.
  Arms: 50 millions AdMSC dose
Drug: CellREADY® drug product IV dose of 100 millions — Allogeneic AdMSC (CellREADY® drug product), intravenous administration, dose of 100 millions.
  Initially, 3 patients will receive the lowest dose (50x106 AdMSC). If the safety analysis of the first 3 patients infused at dose 50x106 AdMSC does not show clinically significant AEs after 6 months of follow-up, 100x106 AdMSC administration may be started in 3 new patients. On the other hand, if safety analysis of the first 3 patients shows a clinically significant AE, 3 new patients will be injected at this same dose before making a final decision on the possibility of dose escalation. Thus, the "100x106 AdMSC " group will only start after the 6-month follow-up and safety analysis completed in the "50x106 AdMSC " group. For each dose, all patients will be followed for 6 months post-injection with 6 visits.
  Arms: 100 millions AdMSc dose
Diagnostic Test: cerebral RMI — cerebral RMI at V1, V5 and V6
Diagnostic Test: PET scan — amyloïde PET scan (flutémétamol) at V1 and V6

SUMMARY:
A3D is a phase I/II clinical trial. The primary objective is to evaluate the safety of allogeneic adipose tissue derived-stem cells (AdMSC) administered by intravenous (IV) route in mild to moderate Alzheimer disease (AD) using a dose escalation protocol.

DETAILED DESCRIPTION:
Bone narrow derived-stem cells (MSC) or adipose tissue-derived stem cells (AdMSC) are widely used in clinical research. The allogeneic approach is currently being considered in indications such as Crohn's disease and graft-versus-host disease. The potential effects of MSCs would be associated with paracrine effects via the secretion of neurotrophic cytokines capable of stimulating endogenous neurogenesis, anti-inflammatory, and immuno-modulatory factors. The recent CRATUS study consisting of IV administration of allogeneic MSCs in frail elderly participants showed a positive effect on functional performance, cognitive performance and inflammation measures. A3D is a phase I/II clinical trial whose primary objective is to evaluate the safety of allogeneic AdMSC IV administration in mild to moderate AD using a dose escalation protocol. Initially, 3 patients will receive the lowest dose (50x106 AdMSC). If the safety analysis of the first 3 patients injected by 50x106 AdMSC does not show clinically significant adverse events (AE) after 6 months of evaluation, 100x106 AdMSC administration may be started in 3 new patients. On the other hand, if the safety analysis of the first 3 patients shows a clinically significant AE related to the treatment, 3 new patients will be infused at this same dose before making a final decision on the possibility of dose escalation. Thus, the "100x106 AdMSC " group will only start after the 6-month follow-up and safety analysis completed in the "50x106 AdMSC " group.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 50 and 85 years old
* AD diagnosis according to NIA-AA 2011 criteria at a mild to moderate stage :

MMSE score between 14 and 26 (include) positive AD amyloid biomarker

* CDR (clinical dementia rating) score ≥ 1
* Patient with no absolute contraindications for PET or MRI scans
* Consent signed by the patient and study partner
* presence of primary caregiver
* Patient with social security coverage

Exclusion Criteria:

* Brain disease (other than AD) that may cause dementia
* Presence of concomitant pathologies not permitting participation in the study
* Concurrent participation in other research that may influence the testing of the A3D study
* Carrier of a pacemaker, valve prosthesis or other internal magnetic or electronic system, history of neurosurgery or aneurysm surgery, presence of metal fragments in the eyes, brain or marrow, claustrophobia
* PET scan performed in the previous year (research context)
* History of cancer diagnosed within the last 5 years
* Presence of > 4 brain microbleeds, a single area of superficial siderosis, or evidence of previous macrohaemorrhage assessed by brain MRI scan
* Regular use of corticosteroids or other steroidal anti-inflammatory drugs (e. g. prednisone)
* Presence of an autoimmune disease (e. g. rheumatoid arthritis, systemic lupus erythematosus) with the exception of psoriasis
* Pregnant or breastfeeding woman
* Adults under guardianship or other legal protection, deprived of their liberty by judicial or administrative decision For patients who will participate in the optional adipose puncture (only carried out in the Toulouse center): Antithrombotic treatment and xylocaine allergy are prohibited.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
number of participants in each group with a clinically significant serious or non-serious AE related to treatment | 6 months
  The primary outcome is the number of participants in each group with a clinically significant serious or non-serious AE related to treatment. Each AE report should include a description of the event, an assessment of its severity, duration, severity, and causality with IV administration of AdMSC. The occurrence of an AE will be assessed by clinical (at selection visit, injection visit, 1 week, 1 month, 3 months, and 6 months), biological (at selection visit, injection visit, 1 week, 1 month, 3 months, and 6 months) and neuroimaging exams (at selection visit, 3 months, and 6 months).

SECONDARY OUTCOMES:
determination of measures related to immunomodulatory activity (composite outcome) | 6 months
  Measures related to immunomodulatory activity: inflammatory (IL-1β, IL-6, TGF-β1, TNF-α, CRP, D-Dimers) and anti-inflammatory (IL-10) blood markers. Markers derived from brain MRI scan (Magnetic resonance sequence Spectroscopy MRS, in the posterior cingulate region, myo-inositol). Immunomonitoring with evaluation of activated T lymphocytes (CD3/CD25/CD69).
determination of measures related to cerebral amyloid load (composite outcome) | 6 months
  Measures related to cerebral amyloid load: The global standardized relative Uptake Value ratio (SUVr) and by regions of interest (anterior cingulum, posterior cingulum, temporal, parietal, precuneus, frontal) assessed by amyloid PET scan (flutémétamol).
determination of measures related to neurotrophic activity (composite outcome) | 6 months
  Cortical thickness assessed by brain MRI scan (T1 weighted sequence). Blood light chain neurofilaments. N-AcetylAspartate by MRS (posterior cingulum)

CONTACTS AND LOCATIONS:
Overall Officials: Julien DELRIEU, MD_PH, Principal Investigator — University Hospital of Toulouse